CLINICAL TRIAL: NCT02340702
Title: COPD in Patients Hospitalized for Acute Decompensated Heart Failure.
Brief Title: Chronic Obstructive Pulmonary Disease (COPD) in Patients Hospitalized for Acute Decompensated Heart Failure.
Acronym: COPD
Status: Withdrawn | Type: Observational
Why Stopped: Unable to abstract pulmonary function and some other data from medical records.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mohammed Yousufuddin, M.D, PI, Mayo Clinic
Other Study IDs: 14-006196
Record Dates: First submitted 2015-01-07; First posted 2015-01-19 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Disease
Keywords: COPD and heart failure
MeSH Terms: conditions — Disease; Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with COPD and those without COPD: The participants of acute decompensated heart failure national registry would be stratified in to two group: those with COPD and those without COPD, to determine prognostic implication of COPD in participants with acute decompensated heart failure
  Interventions: Other: COPD

INTERVENTIONS:
Other: COPD — COPD as diagnosed clinically or based on pulmonary function test showing post-bronchodilator forced expiratory volume in one second to forced vital capacity ratio of <0.7.
  Other Names: chronic obstructive pulmonary disease

SUMMARY:
The presence of chronic obstructive pulmonary disease (COPD) would confer increased in-hospital mortality and length of hospital stay in patients with acute decompensated heart failure Assess the (1) prevalence of COPD in patients who are hospitalized for acute decompensated heart failure and (2) the association between COPD and in-hospital mortality or length of stay in this cohort.

DETAILED DESCRIPTION:
Background:

The prevalence of mild to moderate COPD is ~5%-10% with one-year mortality around 3% while heart failure affects is1%-3% with one year mortality 5-7% in the community. The mortality of COPD and heart failure dramatically increase following hospitalization.

Heart failure and COPD are independent predictors of increased morbidity and mortality. COPD and heart failure frequently co-exist in an individual patient through the shared risk factors. The prevalence of COPD in heart failure patient-population and vice verse varies widely according to patient-selection and age of the population. Estimates suggest that COPD is present in 10-40% of the patients with heart failure. Conversely, unrecognized heart failure is identified in approximately 20% of the patient with COPD. The impact of COPD on clinical outcome in patients with acute decompensated heart failure is unclear.

Methods:

This is an observational cohort study. Per national registry, acute heart failure is defined as either new onset heart failure or decompensation of chronic established heart failure with symptoms sufficient to warrant hospitalization.

The data related to the following variables would be collected:

age, gender, severity of heart failure (mild, moderate, and severe prior to admission), presence of dyspnea, peripheral edema, crackles, systolic and diastolic blood pressure (on admission and on discharge), heart rate (on admission and on discharge), oxygen saturation (on admission and discharge), blood urea nitrogen (on admission and discharge), serum creatinine (on admission and discharge), serum sodium (on admission and discharge), hemoglobin (on admission and discharge), red cell distribution width (on admission and discharge), electrocardiographic intervals (on admission and discharge), comorbidities (coronary artery disease, chronic kidney disease, atrial fibrillation, diabetes, hypertension, dyslipidemia, peripheral artery disease, COPD/asthma, left ventricular ejection fraction >40%. Medication use: angiotensin converting enzyme inhibitors, angiotensin receptor blockers, aspirin, metoprolol tartrate, metoprolol succinate, carvedilol, atenolol, amlodipine, Cardizem, clopidogrel, digoxin, diuretics, statins, nitrates, warfarin, non-steroidal anti-inflammatory drugs, hydralazine.

End-points:

1) All cause in-hospital death and 2) length of hospital stay between heart failure patients with COPD and those with no COPD.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure

Exclusion Criteria:

* Ambulatory patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for acute decompensated heart Failure
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | Average of 5-weeks
  Participants would be followed for the duration of hospital stay

SECONDARY OUTCOMES:
Length of hospital stay | Average of 5-weeks

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials